CLINICAL TRIAL: NCT06605820
Title: Shared Decision-making and Antimicrobial Stewardship in Secondary Care: Exploring Opportunities Along the Start Smart Then Focus Patient Pathway
Brief Title: Shared Decision-making and Antimicrobial Stewardship in Secondary Care
Acronym: SHARE
Status: Recruiting | Type: Observational
Sponsor: Royal Cornwall Hospitals Trust (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 2023.RCHT.05
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Antibiotic Prescribing is the Study Focus (no Condition)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Other: None - Interview Only
- Healthcare workers
  Interventions: Other: None - Interview Only

INTERVENTIONS:
Other: None - Interview Only — None - Interview Only

SUMMARY:
To identify opportunities for antibiotic prescribing shared decision making between patients and prescribers in secondary care.

DETAILED DESCRIPTION:
This is a qualitative study with patients and clinicians in secondary care.

We will use semi-structured interviews with patients and clinicians to address the research question. Patients that have received antibiotics during a recent inpatient stay will be identified using the hospital electronic prescribing system and a letter inviting study participation will be included in their discharge medication pack. Senior prescribing decision makers will be recruited from participating hospitals. In total, we hope to carry out up to 50 interviews with patients and clinicians.

ELIGIBILITY:
Inclusion Criteria:

For clinicians:

* Participant is willing and able to give informed consent for participation in the study.
* Senior registrar or consultant medical or surgical doctor working at participating hospitals and caring for inpatients.
* Fluent in English.

For patients:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 16 years or above (no upper age limit).
* Good standard of speaking English and able to read and understand study materials.
* Received antibiotic for treatment of suspected or confirmed bacterial infection during inpatient stay.

Exclusion Criteria:

* For clinicians:

  * Prescribers not currently caring for inpatients

For patients:

• Patient who received prophylaxis antibiotics only

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will use semi-structured interviews with patients and clinicians to address the research question. Patients that have received antibiotics during a recent inpatient stay will be identified using the hospital electronic prescribing system and a letter inviting study participation will be included in their discharge medication pack. Senior prescribing decision makers will be recruited from participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Patient and prescriber views and experiences with shared decision making (SDM) around antibiotic prescribing in secondary care and to identify further opportunities for SDM. | 1 year
  Data will be analysed using thematic analysis

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Chelsea and Westminster Hospital, Truro